CLINICAL TRIAL: NCT04713150
Title: HEALthy Brain and Child Development Study - COVID-19 Supplement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Charles Alexander Nelson III, Principle Investigator, Boston Children's Hospital
Other Study IDs: P00035929
Record Dates: First submitted 2020-12-17; First posted 2021-01-19 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Child Development; Prenatal Infection; Prenatal Stress; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Positive During Pregnancy: Sixty mother-child dyads, who have or had a confirmed positive COVID-19 test during pregnancy, will be recruited and enrolled in this study. All women enrolled must be 18 years of age or older. Her child will go on to participate at 2-5 days of age, and again at 3-, 6-, 9-, 12- and 24-months of age.
  Interventions: Other: No Intervention
- COVID-19 Negative During Pregnancy: Twenty-five mother-child dyads, who have a confirmed negative COVID-19 test during pregnancy will be recruited and enrolled in the study. Women without any SARS-CoV-2 positive test during pregnancy or any suspected COVID illness, even if not tested, will be enrolled. All women enrolled must be 18 years of age or older. Her child will go on to participate at 3-, 6-, 9-, 12- and 24-months of age.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
The purpose of this study is to advance the scientific understanding of how a prenatal COVID-19 infection and associated psychological distress influences infant neurodevelopment. This project will aim to shed light on how families and child development are impacted by the current COVID-19 pandemic and will work to better support these families and children as they grow.

DETAILED DESCRIPTION:
Prenatal exposure to maternal illness and stress has been widely associated with adverse neurodevelopmental outcomes, including deficits in cognition and socioemotional development. The principal goal of this project utilizes Magnetic Resonance Imaging (MRI), Electroencephalography (EEG), and a variety of behavioral measures to assess brain maturation and neurodevelopment among infants exposed prenatally to COVID-19 and associated high levels of stress. The planned experiments are effective in identifying brain markers that may contribute to resiliency in young infants, determining measures of stress response in relation to a maternal COVID-19 diagnosis, and characterizing the neurodevelopment of those infants born to mothers with a COVID-19 infection.

Specific goals include:

1. To determine the prevalence of psychological distress in pregnant women with a confirmed COVID-19 diagnosis and to examine the extent to which existing high risk environments play a role in the susceptibility of heightened psychological distress.
2. To examine the effects of prenatal distress and maternal illness/inflammation related to a maternal COVID-19 diagnosis on early structural and functional brain development.
3. To characterize neural networks that may have been impacted by a maternal COVID-19 infection and related stress during pregnancy.
4. To assess the early neurodevelopment outcomes of infants exposed to elevated prenatal stress related to a maternal COVID-19 diagnosis during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish- speaking of any ethnicity
* Women, aged 18 or older
* Women who received COVID-19 diagnoses during pregnancy OR Women without any SARS-CoV-2 positive test during pregnancy, any suspected COVID illness (even if not tested) or who received a negative COVID-19 test result during pregnancy

Exclusion Criteria:

Participants will be excluded if the child:

* is born at less than 34 weeks or if birth weight is not appropriate for dates
* has an identified genetic, metabolic, syndromic or progressive neurological disorder (e.g., Down Syndrome, Rett Syndrome, Tuberous Sclerosis, Neurofibromatosis, Fragile X Syndrome) at birth or within the first year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Infants born to COVID-19-positive and COVID-19-negative women.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Maternal stress associated with a SARS-CoV-2 diagnosis in pregnancy. | 9 months (Third trimester - 6 month postnatal visit)
  Using the Perceived Stress Scale (scores can range from 0 to 40, with higher scores indicating greater stress).
Maternal mental health associated with a SARS-CoV-2 diagnosis in pregnancy. | 30 months (Third trimester - 24 month postnatal visit)
  Using the Edinburgh Postnatal Depression Scale (scores range from 0-30, with higher scores indicating greater feelings of depression).
Inventory of maternal experience associated with a SARS-CoV-2 diagnosis in pregnancy. | 30 months (Third trimester - 24 month postnatal visit)
  Using the Recent Life Events Questionnaire (indexes 30 common life events that encompass both positive and negative events).
Inventory of maternal experience related to healthcare associated with a SARS-CoV-2 diagnosis in pregnancy. | 30 months (Third trimester - 24 month postnatal visit)
  Using the COPE Survey (50-item inventory of experiences for new or expectant mothers during the COVID-19 pandemic; psychometric properties and scoring procedures for this measure have yet to be determined).
Global cognitive ability of offspring | 3 months, 6 months, 9 months, 12 months, and 24 months
  Using the Mullen Scales of Early Learning at 3 months and 6 months postnatally. Five skill areas are measured: Gross Motor and four cognitive skills. These cognitive skill are summarized into an Early Learning Composite (scores are permitted to range from 20 to 80) - Fine Motor, Visual Reception, Receptive Language, and Expressive Language. The raw scores for each scale can be converted into age-adjusted normalized scores.
Neural networks of offspring | 3 months, 6 months, 9 months, 12 months, and 24 months
  Using Electroencephalography at 3 months and 6 months postnatally
Early structural and functional brain development of offspring | 1-2 days of life and/or 3-9 months of life
  Using MRI imaging, which will be obtained at 1-2 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Nelson, PhD, Principal Investigator — Boston Children's Hospital
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Laboratories of Cognitive Neuroscience, Boston Children's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided